CLINICAL TRIAL: NCT01249924
Title: The Effectiveness of Perioperative CPAP to Reduce the Occurrence of Sleep Apnea Related Adverse Events in Surgical Patients With Obstructive Sleep Apnea
Brief Title: The Effectiveness of Perioperative CPAP to Reduce Obstructive Sleep Apnea Related Adverse Events
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Dr. Frances Chung, Anesthesiologist, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0000
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2012-07

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: Obstructive sleep apnea (OSA), continuous positive airway pressure(CPAP), surgery, anesthesia
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP Group (Other): CPAP Treatment
  Interventions: Device: auto-titrated CPAP
- Control Group (Other): Routine care
  Interventions: Device: auto-titrated CPAP; Device: Control

INTERVENTIONS:
Device: auto-titrated CPAP — Patients will be treated with auto-CPAP preoperatively for 2-3 nights preoperatively and 5 nights postoperatively during their sleep.
Device: Control — Patients in this group will receive routine care, undergo sleep study on the third postoperative night and be monitored by a pulse oximeter for oxygen saturation level for 2-3 nights preoperatively and 5 nights postoperatively during their sleep.
  Arms: Control Group

SUMMARY:
Objective of the study: To determine whether Perioperative Auto-CPAP treatment prevent postoperative worsening of OSA and improve nocturnal oxygen saturation in surgical patients with moderate and severe OSA.

DETAILED DESCRIPTION:
The patients will be approached by the study coordinators at the preoperative clinic. If the patient is interested in participating the study, STOP-Bang and Epworth questionnaires will be implemented to determine the risk for OSA.If the patients are classified as high risk of having OSA, they are scheduled for an overnight sleep study at home. The patients with Apnea-Hypopnea Index (AHI)>15 from the sleep study will be randomized into two study groups: Perioperative CPAP group or control group (routine care). In the perioperative CPAP group, patients will be treated with auto-CPAP for 2-3 nights preoperatively and 5 nights postoperatively. All patients will undergo sleep study on the third postoperative night and be monitored by a pulse oximeter for 2-3 nights preoperatively and 5 nights postoperatively.

ELIGIBILITY:
Inclusion Criteria:

the patients who meet the following criteria will be recruited

* Patients who are scheduled for inpatient surgery that required a minimum of three nights of hospital stay
* Age: >18 and <80 years old.
* Identified as high risk of having OSA or diagnosed with OSA without using CPAP.

Exclusion Criteria:

* Undergoing nasal, eye, head/neck surgery, intracranial or cardiac/thoracic surgery.
* Unwilling or unable to give informed consent.
* Currently undergoing treatment for sleep apnea including CPAP.
* Requiring prolonged postoperative ventilation.
* New York Heart Association functional class III and IV.
* Having valvular heart disease, dilated cardiomyopathy, implanted cardiac pacemaker, or unstable angina.
* Having myocardial infarction or cardiac surgery within 3 months.
* Having chronic obstructive pulmonary disease, or asthma.
* Having a presence of tracheostomy, facial, neck, or chest wall abnormalities.
* Having abdominal aortic aneurysm surgery, chemotherapy, or immunosuppressive therapy within 3 months.
* Visiting preoperative clinic less than 3 days before scheduled surgery date.
* On nasogastric tube postoperatively.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index | On the third night after surgery
  Apnea-hypopnea index.

SECONDARY OUTCOMES:
Nocturnal oxygen desaturation index (ODI) and percentage of time with SaO2<90%(CT90) | 2-3 nights before surgery and 5 nights after surgery
  Nocturnal oxygen desaturation index (ODI) and percentage of time with SaO2<90%(CT90).

CONTACTS AND LOCATIONS:
Overall Officials: Frances Chung, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Toronto Western Hospital, Department of Aneshtesia, Toronto, Ontario
  - Mount Sinai Hospital, Department of Anesthesia, Toronto, Ontario